CLINICAL TRIAL: NCT00906906
Title: Validation of Venous Cannulae Flow Ratings of the DLP Right Angle Cannulaes Utilizing Ultrasound Transit Time Technology
Brief Title: Validation of Venous Cannulae Flow Ratings
Status: Withdrawn | Type: Observational
Why Stopped: No patient has been enrolled in this study for more than 8 years. Study is closed.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Sponsor
Other Study IDs: 122007-025
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient to receive CPB
  Interventions: Device: Doppler probes

INTERVENTIONS:
Device: Doppler probes — Probes to be placed on CPB tubing to measure blood flow

SUMMARY:
The purpose of this study is to characterize blood flow in the plastic tubing of a heart-lung bypass machine during heart surgery. Technical specifications provided by the manufacturer do not consider varying hemodynamic conditions such as temperature and hemoglobin levels which affect blood viscosity and ultimately blood flow to and from the patient during heart-lung bypass.

The investigator wishes to perform a prospective study of the heart-lung bypass tubing in children that require heart-lung bypass during heart surgery.

DETAILED DESCRIPTION:
During bypass, venous drainage is essential for maintaining proper perfusion of a pediatric patient. The quality of venous drainage has a large impact on the level of care the patient is provided. This study will investigate blood flow velocities through right angle venous cannulae which are utilized during bypass. The flows from each cannulae will be analyzed by using doppler flow probes which employ Transit Time Technology. This type of technology has crystals within the flow probes which send magnetic signals through the tubing with the purpose to determine the most accurate flows of blood. There is little evidence that identifies the actual amount of blood flow generated from each venous cannulae in a clinical setting. Manufacturers of venous cannulae for CPB publish flow ratings for the different sized cannulae available. These flow ratings are gathered from data produced in a non-clinical lab and are often very inaccurate. Because of this inaccuracy, selection is based on experience rather than published clinical data. This study would be instrumental in determining any and all potential risks or benefits to the patient as a result of the amount of drainage provided by the venous cannulae during bypass. A sample size of 50 patients (n=50) over one day old will be utilized for this study. The specific venous cannulae sizes that will be analyzed are the 12Fr, 14Fr, 16Fr, 18Fr, 20Fr, 24Fr, & 28Fr DLP (DLP and Fr are the type and size of cannulae, respectively) right angle cannulae. The doppler flow probes that will be utilized during this study are reusable, non-invasive, clamp-on devices which measure blood flow through the CPB tubing. Each patient will have one flow probe placed on each venous cannulae prior to starting CPB. Bypass itself will not be altered in anyway. Hemoglobin blood levels, blood temperature, and pressure from the venous line will be recorded throughout CPB and are digitally sampled via the CPB machine (e.g. no blood draw required). To further examine the quality of venous drainage, a pressure transducer will be attached to the venous line measuring the amount of negative pressure being generated by the venous cannulae. The negative pressure line will be attached to the venous line at a stopcock that is already present in our CPB circuit. Each cannulae size will be analyzed three times to acquire the proper amount of data needed to fulfill the statistical and practical needs for the study. A descriptive analysis of the continuous and categorical data will be performed using means, standard deviations, confidence intervals, proportions, and frequency distributions. Statistical testing will include parametric and non-parametric bi-variate and multi-variate techniques as appropriate to the variables' level of measurement and distributions.

Notes: 1/15/2025 -Record transferred from Ann & Robert H Lurie Children's Hospital of Chicago to University of Texas Southwestern Medical Center since Record shows UTSW as the Sponsor. Dr. Forbess (Responsible Party) and his team for this study no longer at UTSW to shed light on why this record was transferred to Lurie Children's in 2019. Dr. Jaquiss from Cardiovascular & Thoracic Surgery Department at UTSW confirmed on 1/7/2025 that - "No patient has been enrolled in this study and should be considered to be closed".

ELIGIBILITY:
Inclusion Criteria:

* All Patients that require cardiopulmonary bypass during cardiac surgery.

Exclusion Criteria:

* The only exclusion criteria would be if CPB is not required for surgical repair.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who undergo heart-lung bypass during surgical correction of their congenital or acquired heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12-01 (Actual); Study Completion 2009-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ginther, CCP, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States